CLINICAL TRIAL: NCT02418338
Title: Evaluation of Myocardial Function by Two Dimensional Speckle Tracking Echocardiography in Children With Duchenne Muscular Dystrophy Versus Healthy Children: a Comparative Transversal Multicenter Study
Brief Title: 2D Strain Evaluation: Children With Duchenne Muscular Dystrophy Versus Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9458
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dmd children (Experimental): echocardiography
  Interventions: Other: speckle tracking (2D strain) echocardiography
- healthy children (Other): echocardiography
  Interventions: Other: speckle tracking (2D strain) echocardiography

INTERVENTIONS:
Other: speckle tracking (2D strain) echocardiography — 2D echocardiography videos of both ventricles to perform 2D strain post-examination evaluation

SUMMARY:
Compare systolic function of left ventricle (LV) and right ventricle (VD) by 2D strain evaluation in Duchenne muscular dystrophy children versus a control group.

DETAILED DESCRIPTION:
Among the new echocardiographic techniques, two dimensional Speckle Tracking Imaging or "2D Strain" allows a dynamic study of regionalized and global ventricular contraction. With software for the spatial and temporal processing of a standard 2D image, this technique measures the displacement of natural markers present on the myocardial wall.

Used in adult cardiology since 2000, it could be eligible to pediatric population because of many potential applications. In Duchenne muscular dystrophy, myocardial disease leads to death in the third decade. Early diagnosis and preventive therapy remain a challenge. No clinic, biologic or radiologic markers can predict myocardial disease before advanced and irreversible heart failure.

Recent animals and human studies suggest that 2D strain anomalies could predict left ventricular systolic dysfunction in Duchenne muscular dystrophy. If it is confirmed, 2D strain could be used as early marker of myocardial disease in routine patient follow-up and in future therapeutic studies.

Purpose : - To compare systolic function of left ventricle (LV) and right ventricle (RV) by 2D strain evaluation in Duchenne muscular dystrophy children versus a control group.

* To correlate 2D Strain variables to conventional LV and RV echo variables.
* To evaluate 2D strain feasibility in normal children and Duchenne muscular myopathy population

ELIGIBILITY:
Inclusion Criteria:

* Duchenne's muscular dystrophy (group 1) followed in our institution's referral center of neuromuscular diseases, during regular annual echocardiography follow-up.
* Healthy children (group 2), addressed in pediatric cardiology

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2014-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
global longitudinal LV 2D strain | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, PhD, Principal Investigator — UH Montpellier; Pierre MP Meyer, MD, PhD, Principal Investigator — UH Montpellier; Arnaud BERTRAND, MD, PhD, Principal Investigator — UH Montpellier; Jean-Michel RAUZIER, MD, PhD, Principal Investigator — UH Nîmes; Charlène BREDY, MD, PhD, Principal Investigator — UH Montpellier; François RIVIER, MD, PhD, Principal Investigator — UH Montpellier; Grégoire DE LA VILLEON, MD, PhD, Principal Investigator — UH Montpellier; Ulrike WALTHER-LOUVIER, MD, PhD, Principal Investigator — UH Montpellier; Sophie GUILLAUMONT, MD, PhD, Principal Investigator — UH Montpellier; Camille SOULATGES, MD, PhD, Principal Investigator — UH Montpellier; Marie VINCENTI, MD, PhD, Principal Investigator — UH Montpellier
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

REFERENCES:
- [Background] Amedro P, Vincenti M, De La Villeon G, Lavastre K, Barrea C, Guillaumont S, Bredy C, Gamon L, Meli AC, Cazorla O, Fauconnier J, Meyer P, Rivier F, Adda J, Mura T, Lacampagne A. Speckle-Tracking Echocardiography in Children With Duchenne Muscular Dystrophy: A Prospective Multicenter Controlled Cross-Sectional Study. J Am Soc Echocardiogr. 2019 Mar;32(3):412-422. doi: 10.1016/j.echo.2018.10.017. Epub 2019 Jan 21. PMID 30679141
- [Derived] Lanot N, Vincenti M, Abassi H, Bredy C, Agullo A, Gamon L, Mura T, Lavastre K, De La Villeon G, Barrea C, Meyer P, Rivier F, Meli AC, Fauconnier J, Cazorla O, Lacampagne A, Amedro P. Assessment of left ventricular dyssynchrony by speckle tracking echocardiography in children with duchenne muscular dystrophy. Int J Cardiovasc Imaging. 2022 Jan;38(1):79-89. doi: 10.1007/s10554-021-02369-y. Epub 2021 Dec 14. PMID 34905152